CLINICAL TRIAL: NCT02754128
Title: Linking Neuroplasticity With the Outcomes of Walking-based Interventions: A Feasibility Trial Comparing a Motor Learning Versus a Strength-based Program in Children With Cerebral Palsy
Brief Title: BeFAST or BeSTRONG: Brain Change After Fun Athletic Sports-skill Training or Brain Change After Strength TRaining Focusing ON Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: The Hospital for Sick Children (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-624
Record Dates: First submitted 2016-04-06; First posted 2016-04-28 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2017-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BeFAST (Active Comparator): Motor learning-based program involving athletic lower extremity training of gait-related skills.
  Interventions: Behavioral: BeFAST
- BeSTRONG (Active Comparator): Lower limb strength training program involving progressive muscle resistance exercises.
  Interventions: Behavioral: BeSTRONG

INTERVENTIONS:
Behavioral: BeFAST — The motor learning (ML)-based gait-related training program is designed to improve advanced gross motor skills and athleticism. It will involve 45-min sessions twice to three times weekly over 6 weeks for a total of 16 active sessions. A maximum of 7 weeks will be permitted. Each session will consist of 35-min of active training along with a 10-min active warm-up/cool-down that incorporates ML. Children will be given a 3- to 5-min mental motor imagery script to practice on days when they do not have active training sessions. The total number of sessions (combined training/home imagery) will be five per week.
  Arms: BeFAST
Behavioral: BeSTRONG — The functional strength training program is designed to improve gait-related skills. It will involve 45-min sessions twice to three times weekly over 6 weeks for a total of 16 active sessions. A maximum of 7 weeks will be permitted. Each session will consist of 35-min of active training along with a 10-min active warm-up/cool-down. Children will be given a 3- to 5-min home program of strength exercises to practice on days when they do not have active training sessions. The total number of sessions (combined training/home program) will be five per week.
  Arms: BeSTRONG

SUMMARY:
The purpose of this study is to compare a motor learning (ML)-based gait-related training intervention to a functional lower limb strength training intervention, with a concurrent evaluation of functional, neural and participation outcomes for children and youth with Cerebral Palsy (CP).

This study is a two-group, parallel arm RCT in which twenty-two children with CP in GMFCS Levels I-II will be randomly allocated to a 6-week, 16 session program of: (i) ML based gait training or (ii) lower limb strength training. Outcome assessments occur pre/post/4-months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* 7-17 years old
* diagnosis of hemiplegic or diplegic Cerebral Palsy
* GMFCS Level I-II
* able to follow testing and motor imagery instructions
* able to actively participate in a minimum of 45 minutes (min) of physical activity
* show evidence of independent dorsiflexion of both ankles
* able to commit to attendance of sessions two to three times weekly for six weeks.

Exclusion Criteria:

* orthopaedic surgery within the last 9 months (muscle) or 12 months (bone)
* Botulinum toxin-A (BTX-A) injections to lower limb in the last 4 months
* inability to put BTX-A on hold during trial
* severe spasticity (may be a contraindication for neuroimaging procedures)
* seizure disorder (if not fully controlled by medication for 12 months)
* not prepared or unable to discontinue any formal lower limb therapy intervention or physical activity program during the trial
* involved in another intervention study
* standard MRI contraindications (e.g., magnetic implants, inability to lay still, claustrophobia etc.)

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in advanced motor skills on the Challenge Module | 7 days pre/7 days post/4-months post training intervention
  The Challenge Module is a new published measure of advanced motor skills.

SECONDARY OUTCOMES:
Change from baseline in functional activity in lower-limb related cortical areas, assessed using functional MRI (fMRI) | 7 days pre/7 days post training intervention
Change from baseline in resting state activity, assessed using resting state fMRI | 7 days pre/7 days post training intervention
Change from baseline in microstructure of brain, assessed using diffusion tensor imaging (DTI) | 7 days pre/7 days post training intervention
Change from baseline in Physical Activity self-efficacy | 7 days pre/7days post/4-months post training intervention
  Participant-report measure of Task efficacy and Barrier efficacy for physical activity.
Change from baseline in walking activity, assessed using an Actigraph accelerometer | 7 days pre/7days post/4-months post training intervention
Change from baseline in gait kinematics as measured using an electronic walkway | 7 days pre/7days post/4-months post training intervention
  Time/distance parameters of footsteps via GAITRite system.
Change from baseline in physical activity participation, as measured using the Participation and Environment Measure for Children/Youth (PEM-CY) | 7 days pre/7days post/4-months post training intervention
  Parent-report measure of participation in the home, school and community, as well as environmental factors within each setting.
Change from baseline in walk speed on the Six-minute walk test | 7 days pre/7days post/4-months post training intervention
  Standardized 6 minute walk test (with shoes, orthoses as required) to determine distance covered (capability measure). Well-validated in pediatric CP.
Change from baseline in targeted goal abilities and satisfaction with performance as measured by the Canadian Occupational Performance Measure | 7 days pre/7days post/4-months post training intervention
  Three to five individualized walking-based activity/participation set at baseline with assessor and child/parent, and re-evaluated by child/parent at post-intervention assessments
Change from baseline in targeted goal abilities as measured by Goal Attainment Scaling (GAS) | 7 days pre/7days post/4-months post training intervention
  Three to five individualized walking-based activity/participation set at baseline with assessor and child/parent, and re-evaluated by child/parent at post-intervention assessments

OTHER OUTCOMES:
Motor learning as evaluated using retention and transfer tests | Week 2, 4, 6
  Individualized skills will be identified to practice at every session (retention) and only at sessions 5/10/15 (transfer) to evaluate motor learning
Motor learning content of interventions, as assessed using the Motor Learning Strategy Rating Instrument (MLSRI) | Week 2, 4, 6
  The MLSRI is used to assess the extent to which motor learning strategies are used within an intervention session
Intervention program enjoyment, assessed using a modified version of the Physical Activity Enjoyment Scale (PACES) | 7 days post training intervention
  Participants' enjoyment of the intervention program will be assessed following the intervention
Intervention session enjoyment | 16 times over 6 weeks (following each intervention session)
  Participants' enjoyment of each session will be assessed using a study-specific questionnaire
Rating of exertion, assessed using Pictorial Children's Effort Rating Table (PCERT) | Completed at 22 minutes (mid-point) and at 43-minutes (2-minutes before end) of each intervention session
  Children will be asked to complete PCERT at mid-point of each session, and 2 minutes before session completion
Heart rate (beats per minute) | Assessed at 4 time points per session: 1 min before start of session, at 22 minutes (mid-point), at 43-minutes (2-min before end), and at 45-minutes (end) of each session
  Heart rate will be monitored by treating staff member via radial pulse.
Body pain | Completed 2 minutes before and 2 minutes after each intervention session
  Use of FACES pain scale and body diagrams to show areas of pain (musculoskeletal and other)
Parent Satisfaction scale | 7 days post training intervention
  Parent's satisfaction and perceived benefit of intervention will be assessed using a study-specific questionnaire
Staff Satisfaction scale | 7 days post training intervention
  Staff satisfaction and perceived benefit of intervention for each child in the study will be assessed using a study-specific questionnaire
Lower limb strength | 7 days pre/7days post/4-months post intervention
  A 30 second lateral step-up test will be used bilaterally to assess functional lower limb strength
Ankle range of motion and dorsiflexion force | 7 days pre/7days post/4-months post intervention
  Passive and active ROM will be assessed using a goniometer
Dorsiflexion force | 7 days pre/7days post/4-months post intervention
  Dorsiflexion force will be assessed using surface electromyography (EMG)
Change from baseline in lower-limb proprioception | 7 days pre/7days post/4-months post intervention
  Lower limb joint-sense position will be assessed using a semi-goniometer (protocol modified from Wingert et al, 2009)
Mental chronometry | 7 days pre/7days post/4-months post intervention
  Participants will be timed while walking a 10-meter distance, and then timed while imagining walking the same distance.
Motor Imagery Questionnaire for Children (MIQ-C) | 7 days pre/7days post/4-months post intervention
  Participant's motor imagery ability will be assessed using the 12-item MIQ-C
Feasibility process indicators: recruitment rate | Through study completion, an average of 6-months
  Recruitment rate: # eligible participants as compared to # screened and # enrolled
Feasibility process indicators: perceived intervention benefit | Through study completion, an average of 6-months
  Perceived intervention benefit calculated as combined child/parent rating
Feasibility process indicators: retention rate | Through study completion, an average of 6-months
  Number of children enrolled as compared to number of children who complete the study
Feasibility resource indicators: adherence rate | Through study completion, an average of 6-months
  Number of sessions completed
Feasibility resource indicators: data collection time | Through study completion, an average of 6-months
  Projected vs actual data collection time
Feasibility resource indicators: data collection completion | Through study completion, an average of 6-months
  Percent missing data
Feasibility management indicators: Intervention fidelity | Through study completion, an average of 6-months
  Within session effort scores
Feasibility management indicators: Intervention fidelity/contamination | Through study completion, an average of 6-months
  Video sessions every 2 weeks to assess session content: (i) STRONG group: 1RM lower limb strength progression; (ii) FAST group: Session content via Motor Learning Strategy Rating Instrument (MLSRI)
Feasibility management indicators: Intervention fidelity | Through study completion, an average of 6-months
  Completion of diaries for motor imagery/strength home practice
Feasibility management indicators: Intervention fidelity/contamination | Through study completion, an average of 6-months
  Log books for PA-participation tracking/management in active intervention and 4 month follow-up
Feasibility management indicators:Treatment administration | Through study completion, an average of 6-months
  PTA/RKin session summary form data
Feasibility management indicators: Acceptability of intervention | Through study completion, an average of 6-months
  Aggregate score of: Parent/staff satisfaction scale, child Physical Activity Enjoyment Scale (PACES), child intervention satisfaction score
Feasibility science indicators | Through study completion, an average of 6-months
  Treatment response
Feasibility science indicators:adverse events | Through study completion, an average of 6-months
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Wright, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hilderley AJ, Wright FV, Taylor MJ, Chen JL, Fehlings D. Functional Neuroplasticity and Motor Skill Change Following Gross Motor Interventions for Children With Diplegic Cerebral Palsy. Neurorehabil Neural Repair. 2023 Jan;37(1):16-26. doi: 10.1177/15459683221143503. Epub 2022 Dec 15. PMID 36524254